CLINICAL TRIAL: NCT03540836
Title: A Phase 1, Randomized, Open-label, Crossover Study to Determine the Relative Bioavailability of Relacorilant Administered as 3×100-mg Softgel Capsules, 3×100 mg Hard Shell Capsules, and 6×50-mg Hard-shell Capsules in Healthy Adult Subjects
Brief Title: A Study to Determine the Relative Bioavailability of Two New Relacorilant Capsule Variants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CORT125134-127
Record Dates: First submitted 2018-05-17; First posted 2018-05-30 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-08

CONDITIONS: Healthy
MeSH Terms: interventions — relacorilant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Relacorilant 3x100mg softgel capsules (Experimental): Relacorilant (3x100 mg softgel capsules)
  Interventions: Drug: Relacorilant (3x100 mg softgel capsules)
- Relacorilant 3x100mg hard-shell capsules (Experimental): Relacorilant (3x100 mg hard-shell capsules)
  Interventions: Drug: Relacorilant (3x100 mg hard-shell capsules)
- Relacorilant 6x50mg hard-shell capsules (Experimental): Relacorilant (6x50mg hard-shell capsules)
  Interventions: Drug: Relacorilant (6x50mg hard-shell capsules)

INTERVENTIONS:
Drug: Relacorilant (3x100 mg softgel capsules) — A single relacorilant 300mg dose (3x100 mg softgel capsules) will be given once on Day 1 of one of three treatment periods.
  Other Names: CORT125134
  Arms: Relacorilant 3x100mg softgel capsules
Drug: Relacorilant (3x100 mg hard-shell capsules) — A single relacorilant 300mg dose (3x100 mg hard-shell capsules) will be given once on Day 1 of one of three treatment periods.
  Other Names: CORT125134
  Arms: Relacorilant 3x100mg hard-shell capsules
Drug: Relacorilant (6x50mg hard-shell capsules) — A single relacorilant 300mg dose (6x50mg hard-shell capsules) will be given once on Day 1 of one of three treatment periods.
  Other Names: CORT125134
  Arms: Relacorilant 6x50mg hard-shell capsules

SUMMARY:
This is an open-label, randomized, 3 treatment, 3-period, 6-sequence, crossover study conducted at a single study center to characterize the relative bioavailability of relacorilant administered as 3×100-mg softgel capsules (Treatment A), 3×100 mg hard-shell capsules (Treatment B), and 6×50-mg hard shell capsules (Treatment C/reference) in healthy, fasted, adult subjects.

Eligible subjects will participate in 3 treatment periods. During each treatment period, subjects will receive a single 300-mg relacorilant dose. An equal number of subjects will be randomized to each of 6 sequences.

DETAILED DESCRIPTION:
This is an open-label, randomized, 3 treatment, 3-period, 6-sequence, crossover study. Eligible subjects will participate in 3 treatment periods. During each treatment period, subjects will receive a single 300-mg relacorilant dose. An equal number of subjects will be randomized to each of 6 sequences (i.e., ABC, BCA, CAB, BAC, ACB, and CBA):

(A) relacorilant single 300 mg dose (3×100-mg softgel capsules) following a minimum 10 hour fast (Test 1) (B) relacorilant single 300 mg dose (3×100-mg hard-shell capsules) following a minimum 10-hour fast (Test 2) (C) relacorilant single 300 mg dose (6×50-mg hard-shell capsules) following a minimum 10 hour fast (Reference) Subjects will be admitted to the Clinical Research Unit (CRU) on the morning of Day -1 of each period following an 8-hour fast for baseline assessments and will remain confined until Day 3 of each period. After dosing in Period 1 and Period 2, subjects will undergo minimum 14 day washouts between doses of study drug. Subjects will then receive the next relacorilant dose in their randomized sequence in Period 2 and Period 3, respectively. Subjects will attend an outpatient Follow-up Visit 14±2 days after the last dose of study drug in Period 3 (or Early Termination Visit).

Blood samples will be collected before dosing and at intervals up to 120 hours after relacorilant dose in Periods 1, 2 and 3.

Safety and tolerability will be monitored using AEs, clinical laboratory evaluations, 12-lead ECG recordings, vital signs, and physical examinations.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand the purpose and risks of the study; willing and able to adhere to scheduled visits, treatment plans, laboratory tests, and other study evaluations and procedures.
* Give written informed consent.
* Be males or nonpregnant, nonlactating females judged to be in good health, based on the results of medical history, physical examination, vital signs, 12-lead ECG, and clinical laboratory findings.
* Have a body mass index (BMI) between 18 and 32 kg/m2, inclusive, and a body weight more than 50 kg (110 pounds).
* Be a nonsmoker. Use of nicotine or nicotine-containing products must be discontinued at least 90 days prior to the first dose of study drug.
* Be willing to comply with study restrictions
* Have suitable veins for multiple venipuncture/cannulation.
* Female subjects must be either of nonchildbearing potential (i.e., postmenopausal or permanently sterilized) or use highly effective contraception with low user-dependency.

  * The only acceptable method of highly effective contraception with low user-dependency is an intrauterine device (IUD). Use of hormonal contraception (by any route, including intrauterine hormone releasing systems) or hormone replacement therapy is NOT acceptable.

Exclusion Criteria:

* Be an employee or immediate family member of the Clinical Research Unit or Corcept.
* Have been previously enrolled in any study of relacorilant.
* Have multiple drug allergies or be allergic to any of the components of relacorilant.
* Have a condition that could be aggravated by glucocorticoid blockade (e.g., asthma, any chronic inflammatory condition).
* Have a history of malabsorption syndrome or previous gastrointestinal surgery, with the exception of appendectomy and cholecystectomy, which could affect drug absorption or metabolism.
* Current, or previous within a 1-year period, alcohol or substance abuse.
* In the 2 calendar months before first study drug administration, have donated/lost blood or plasma in excess of 400 mL.
* In the 30 days before first study drug administration, have participated in another clinical trial of a new chemical entity or a prescription medicine.
* Have a positive test for alcohol or drugs of abuse at screening or first admission.
* Have clinically relevant abnormal findings on vital signs, physical examination, laboratory screening tests, or 12-lead ECG, at screening and/or before first study drug administration, including but not limited to**:

  * QT interval corrected for heart rate (QTc) using Fridericia's equation (QTcF) >450 ms (from mean of 3 supine ECGs, performed at least 2 minutes apart)
  * Stage 2 or higher hypertension (supine/semi-recumbent systolic blood pressure [SBP] >160 mmHg, diastolic blood pressure [DBP] >100 mmHg; based on mean of duplicate values recorded at least 2 minutes apart)
  * Stage 1 hypertension (supine/semi-recumbent SBP 140-160 mmHg, DBP 90-100 mmHg; based on mean of duplicate values recorded at least 2 minutes apart) associated with indication for treatment i.e., evidence of end-organ damage, diabetes, or a 10-year cardiovascular risk, estimated using a standard calculator, (e.g., QRISK2-2016) greater than 20%
  * Estimated glomerular filtration rate <60 mL/minute/1.73 m2, estimated using the Chronic Kidney Disease Epidemiology Collaboration method (Levey 2009)
  * Hypokalemia (potassium below lower limit of normal)
  * Alanine aminotransferase (ALT), aspartate amino transferase (AST), and/or gamma- glutamyl transferase (GGT) >1.5 times the upper limit of normal (ULN)
  * Seropositive for hepatitis B, hepatitis C, or human immunodeficiency (HIV) viruses **For purposes of qualifying any given subject for study participation, out-of-range values may be repeated once.
* Have any medical or social reasons for not participating in the study raised by their primary care physician.
* Have any other condition that might increase the risk to the individual or decrease the chance of obtaining satisfactory data, as assessed by the Investigator.
* Taken any prohibited prior medication within protocol designated timeframes, such as or including any glucocorticoid, strong inducers, inhibitors or substrates of CYP enzymes involved in drug-drug-interactions, hormonal contraception or hormone replacement therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-05-24 (Actual); Primary Completion 2018-07-16 (Actual); Study Completion 2018-07-25 (Actual)

PRIMARY OUTCOMES:
Area under plasma concentration-time curve up to the last quantifiable sample (AUC0-tz) | pre-dose to 120 hours post-dose in Periods 1 -3.
  Ratio of population geometric means (GMR) of AUC0-tz for Test 1 (relacorilant 3×100-mg softgel capsules) and Reference (relacorilant 6×50-mg hard-shell capsules) and for Test 2 (relacorilant 3×100-mg hard-shell capsules) and Reference (relacorilant 6×50-mg hard-shell capsules)

SECONDARY OUTCOMES:
Area under plasma concentration-time curve extrapolated to infinity (AUCinf) | pre-dose to 120 hours post-dose in Periods 1-3
  Ratio of population geometric means (GMR) of AUCinf for Test 1 (relacorilant 3×100-mg softgel capsules) and Reference (relacorilant 6×50-mg hard-shell capsules and for Test 2 (relacorilant 3×100-mg hard-shell capsules) and Reference (relacorilant 6×50-mg hard-shell capsules)
Maximum plasma concentration (Cmax) | pre-dose to 120 hours post-dose in Periods 1-3
  Ratio of population geometric means (GMR) of Cmax for Test 1 (relacorilant 3×100-mg softgel capsules) and Reference (relacorilant 6×50-mg hard-shell capsules) and for Test 2 (relacorilant 3×100-mg hard-shell capsules) and Reference (relacorilant 6×50-mg hard-shell capsules)
Time to Maximum plasma concentration (Tmax) | pre-dose to 120 hours post-dose in Periods 1-3
  Ratio of population geometric means (GMR) of Tmax for Test 1 (relacorilant 3×100-mg softgel capsules) and Reference (relacorilant 6×50-mg hard-shell capsules) and for Test 2 (relacorilant 3×100-mg hard-shell capsules) and Reference relacorilant 6×50-mg hard-shell capsules)
Adverse Events | up to 30 days after the last dose of study drug
  Incidence of treatment emergent adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Ada Lee, MD, Study Director — Corcept Therapeutics
Locations (1):
- Celerion, Tempe, Arizona, United States